CLINICAL TRIAL: NCT02301195
Title: Measuring the Effects of Therapeutic Horseback Riding on School-Age Children and Adolescents With Autism Spectrum Disorders
Brief Title: Trial of Therapeutic Horseback Riding in Children and Adolescents With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 07-1148; 1R01NR012736 (NIH)
Record Dates: First submitted 2014-11-19; First posted 2014-11-25 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Autism Spectrum Disorder; Child Development Disorders, Pervasive
Keywords: Therapeutic Horseback Riding
MeSH Terms: conditions — Autism Spectrum Disorder; Child Development Disorders, Pervasive | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapeutic Horseback Riding (Experimental): Ten-weekly one-hour manualized small group Therapeutic Horseback Riding intervention led by certified THR instructor.THR intervention taught riding and horsemanship skills.
  Interventions: Other: Therapeutic horseback riding
- Barn Activity Intervention (Active Comparator): Ten-weekly one-hour manualized small group Barn Activity Intervention led by THR instructor, teaching horsemanship skills without horses present.
  Interventions: Other: Barn Activity Intervention

INTERVENTIONS:
Other: Therapeutic horseback riding — Inclusion of horses as part of the therapeutic experience
  Other Names: Equine-Assisted Activities and Therapies; Animinal-Assisted Intervention
  Arms: Therapeutic Horseback Riding
Other: Barn Activity Intervention — Equine-focused educational activities in small group setting without horses
  Arms: Barn Activity Intervention

SUMMARY:
This study is being carried out to learn more about the effects of Therapeutic Horseback Riding (THR) for children and adolescents with an autism spectrum disorder (ASD). This treatment is very popular and horseback riding for children and adults with disabilities has been used as a form of therapy in the United States for over forty years. However, very little research has been done to find out whether or not THR is effective as a therapy for children with an ASD. This study is being done to see if THR will improve the agitation behaviors, coordination, and communication skills of children and adolescents with an ASD. This study is also being done to find out if the horse is necessary for children and adolescents with an ASD to improve.

DETAILED DESCRIPTION:
This study expands previous preliminary equine-assisted intervention research, including the authors' 10-week Therapeutic horseback riding (THR) intervention pilot, by evaluating the effectiveness of therapeutic horseback riding (THR) on self-regulation, socialization, communication, adaptive, and motor behaviors in children with autism spectrum disorder (ASD). Method: One hundred and twenty-seven participants (ages 6-16 years) were randomized by nonverbal IQ standard scores (< 85 or > 85) to one of two 10-week small groups: THR intervention; or barn activity (BA) control group without horses. Both interventions used similar methods, and the fidelity of the THR intervention was monitored. Participants were evaluated within one month pre- and post-intervention by raters blind to intervention conditions and caregiver questionnaires. Weekly during the intervention, caregivers rated participants' behaviors during the preceding week.

ELIGIBILITY:
Inclusion Criteria:

* Score ≥ 11 on the irritability and stereotypy subscales of Aberrant Behavior Checklist-Community
* Nonverbal IQ ≥ 40
* Diagnosis of autistic or Asperger's disorder prior to study admission from a psychologist or psychiatrist in the community
* Meets diagnostic cut-off scores for autism spectrum on the Social Communication Questionnaire (SCQ) (> 15) and on the Autism Diagnostic Observation Schedule, Second Edition (ADOS-2)
* Meets DSM-IV-TR criteria for autistic or Asperger's disorder based on diagnostic information gathered for this study from the SCQ, ADOS-2, and Repetitive Behavior Scales-Revised (RBS-R)
* Absence of significant vision, hearing, or motor impairments
* Absence of genetic disorders known to be causative of or potentially resulting in a phenotype similar to autism: Fragile X Syndrome, Landau Kleffner, Rett Syndrome, Childhood Disintegrative Disorder, or tuberous sclerosis, based on screening by clinical staff
* In the event that a family has more than one child diagnosed with autism or Asperger's, only one child per family will be included in the study that meets other study inclusion criteria to maintain independent observation of the participant
* Must have a consistent school-based teacher (vs. a parent who is providing home schooling) willing to complete the ABC-C form twice during the study for each participant, as well as a parent/guardian who is willing to complete the designated outcome parent/guardian report forms during the study

Exclusion Criteria:

* Child has a medical or psychiatric disorder or behavioral issue that would prevent participation
* Child has had no more than 2 hours exposure to EAATs (equine assisted activities and therapies) in the past 6 months and is judged, during the evaluation at Hearts & Horses by the research site coordinator, to not have significant riding experience (an individual with significant riding experience is defined here as one for whom the beginner curriculum would not be appropriately challenging), as the curriculum is designed for beginner riders
* The child has a history of animal abuse or phobia to horses
* Wards of the State

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 209 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2014-06-19 (Actual); Study Completion 2014-06-19 (Actual)

PRIMARY OUTCOMES:
Change in Aberrant Behavior Checklist-Community (Irritability subscale) | One month pre-intervention, weekly for 10 weeks during intervention, and one month post intervention, and 6 months post intervention
  The investigators hypothesize that social communication behaviors will increase and subjects will show a decrease in aberrant behaviors from pre to post THR lesson and over the course of the 10-week intervention, as observed in the brief periods captured (e.g., estimated 4 minutes before and 4 minutes after each THR lesson).

SECONDARY OUTCOMES:
Change in Aberrant Behavior Checklist-Community (Hyperactivity, Lethargy, Stereotypy subscale) | One month pre-intervention, weekly for 10 weeks during intervention, and one month post intervention, and 6 months post intervention
  The investigators hypothesize that social communication behaviors will increase and subjects will show a decrease in aberrant behaviors from pre to post THR lesson and over the course of the 10-week intervention, as observed in the brief periods captured (e.g., estimated 4 minutes before and 4 minutes after each THR lesson).
Change in Social Responsiveness | One month pre-intervention, weekly for 10 weeks during intervention, and one month post intervention, and 6 months post intervention
  Subjects in the THR group will have greater improvements in socialization, as measured by a parent/guardian report form, the Social Responsiveness Scale, than the control group.
Change in Systematic Analysis of Language Transcript | One month pre-intervention, weekly for 10 weeks during intervention, and one month post intervention, and 6 months post intervention
  Subjects in the THR group will have greater improvement on communication, as measured by blinded speech therapist assessment using the Peabody Picture Vocabulary Test and the Systematic Analysis of Language Transcripts
Change in Peabody Picture Vocabulary Test-4 | One month pre-intervention, weekly for 10 weeks during intervention, and one month post intervention, and 6 months post intervention
  Subjects in the THR group will have greater improvement on communication, as measured by blinded speech therapist assessment using the Peabody Picture Vocabulary Test and the Systematic Analysis of Language Transcripts, as well as by parent interview utilizing the Vineland Adaptive Behavior Scales-II communication subscale, than the control group.
Change in Bruininks-Oseretsky Test of Motor Proficiency-2nd Ed. (Short form) | One month pre-intervention, weekly for 10 weeks during intervention, and one month post intervention, and 6 months post intervention
  Subjects in the THR group will have greater improvement on motor functioning (i.e., physical coordination, stability, and motor planning/praxis), as measured by blinded Occupational Therapists assessment utilizing the Bruininks-Oseretsky Test of Motor Proficiency and the Sensory Integration and Praxis Test, than the control group.
Change In Sensory Integration and Praxis Test (Praxis on verbal command & Postural Praxis subtests) | One month pre-intervention, weekly for 10 weeks during intervention, and one month post intervention, and 6 months post intervention
  Subjects in the THR group will have greater improvement on motor functioning (i.e., physical coordination, stability, and motor planning/praxis), as measured by blinded Occupational Therapists assessment utilizing the Bruininks-Oseretsky Test of Motor Proficiency and the Sensory Integration and Praxis Test, than the control group.
Change in Vineland Adaptive Behavior Scales Interview 2nd Ed. | One month pre-intervention, weekly for 10 weeks during intervention, and one month post intervention, and 6 months post intervention
  subjects in the THR group will have statistically non-significant changes in their post-intervention scores on communication, as measured by blinded speech therapist assessment using the Peabody Picture Vocabulary Test and the Systematic Analysis of Language Transcripts, as well as by parent interview utilizing the Vineland Adaptive Behavior Scales-II communication subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Gabriels, PsyD, Principal Investigator — University of Colorado Denver/Children's Hosptial Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petty JD, Pan Z, Dechant B, Gabriels RL. Therapeutic Horseback Riding Crossover Effects of Attachment Behaviors with Family Pets in a Sample of Children with Autism Spectrum Disorder. Int J Environ Res Public Health. 2017 Mar 3;14(3):256. doi: 10.3390/ijerph14030256. PMID 28273822
- [Result] Gabriels RL, Pan Z, Dechant B, Agnew JA, Brim N, Mesibov G. Randomized Controlled Trial of Therapeutic Horseback Riding in Children and Adolescents With Autism Spectrum Disorder. J Am Acad Child Adolesc Psychiatry. 2015 Jul;54(7):541-9. doi: 10.1016/j.jaac.2015.04.007. Epub 2015 May 5. PMID 26088658
- [Derived] Pan Z, Granger DA, Guerin NA, Shoffner A, Gabriels RL. Replication Pilot Trial of Therapeutic Horseback Riding and Cortisol Collection With Children on the Autism Spectrum. Front Vet Sci. 2019 Jan 14;5:312. doi: 10.3389/fvets.2018.00312. eCollection 2018. PMID 30693284
- [Derived] Gabriels RL, Pan Z, Guerin NA, Dechant B, Mesibov G. Long-Term Effect of Therapeutic Horseback Riding in Youth With Autism Spectrum Disorder: A Randomized Trial. Front Vet Sci. 2018 Jul 16;5:156. doi: 10.3389/fvets.2018.00156. eCollection 2018. PMID 30062099
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4475278